CLINICAL TRIAL: NCT02685007
Title: RollOut -Pre-Rolled TachoSil in Laparoscopic Utilisation. A Non-Interventional Study
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TachoSil-4001; NIS005460 (Registry Identifier: AGES)
Record Dates: First submitted 2016-02-08; First posted 2016-02-18 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Laparoscopy
Keywords: minimal invasive surgery
MeSH Terms: interventions — TachoSil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Inpatients: Inpatients planned for laparoscopic surgery, in the field of gynecology, urology and visceral surgery will be documented from of surgery until date of discharge from hospital
  Interventions: Other: Tachosil

INTERVENTIONS:
Other: Tachosil — TachoSil is a collagen matrix that is coated with human fibrinogen and human thrombin.

SUMMARY:
The purpose of this study is to describe ease of use and satisfaction with application of the pre-rolled TachoSil in laparoscopic procedures within approved therapeutic indication as per Summary of Product Characteristics (SmPC).

DETAILED DESCRIPTION:
The drug being observed in this study is called Tachosil. Tachosil is being used in open invasive surgery for use as a local haemostatic and tissue sealing. This study will look at the application and an overview on the ease of use of pre-rolled form of Tachosil in minimal invasive (laparoscopic) surgery, cost analysis along with the evaluation of participant's satisfaction with the product.

The study will enroll approximately 131 participants who will be inpatients. A participant can be included in the study when the physician has decided to use pre-rolled TachoSil according to the local SmPC and after obtaining informed consent from the participant. Participants will be analyzed in a routine setting after surgery.

Data from all participants will be collected from their files as well as study specific questions answered by the treating physician.

This multi-center trial will be conducted in 7 Austrian centers. The overall recruitment period is expected for 1 year and six months. Participants will be analyzed from the date of surgery till their discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

1- Inpatients planned for laparoscopic surgery, in the field of gynecology, urology and abdominal surgery where pre-rolled TachoSil was applied, 18 years or older.

Exclusion Criteria:

1. Has contraindications, such as hypersensitivity to the active pharmaceutical ingredients or to other components of pre-rolled TachoSil according to the current SmPC.
2. Is participating in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include inpatients planned for laparoscopic surgery, in the field of gynecology, urology and visceral surgery and where pre-rolled TachoSil will be applied.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2016-04-05 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (8):
- Austria (8):
  - Landeskrankenhaus Hochsteiermark, Standort Bruck a.d. Mur; Abteilung fur Chirurgie, Bruck an der Mur
  - LKH Universitatsklinikum Graz Universitatklinik fur Chirurgie; Abteilung fur Allgemeinchirurgie, Graz
  - Landeskrankenhaus Hall; Allgemeine Chirurgie, Hall in Tirol
  - Kepler Universitatsklinikum GmbH Med Campus III.; Abteilung Chirurgie II, Linz
  - Krankenhaus der Barmherzigen Schwestern Linz Betriebsges.m.b.H, Linz
  - Landeskrankenhaus Salzburg/SALK Universitatsklinikum der PMU; Univ.-Klinik fur Urologie und Andrologie, Salzburg
  - Univ.-Klinik fur Chirurgie; Klin. Abt. fur Allgemeinchirurgie, Vienna
  - Klinikum Wels-Grieskirchen GmbH; Abteilung fur Urologie, Wels

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in Austria from 05 April 2016 to 14 August 2017.
Pre-assignment Details: Participants planned for laparoscopic surgery in the field of gynecology, urology or visceral surgery were enrolled in this study to use pre-rolled TachoSil according to the local Summary of Product Characteristics (SmPC) based on physician decision and the data was collected under routine standard of care.
Groups:
- TachoSil: TachoSil, sealant matrix coated with fibrinogen and thrombin, epilesional application, applied during surgery in participants who had laparoscopic surgery, in the field of gynecology, urology and visceral surgery according to the local SmPC.
Period: Overall Study
Arm/Group | TachoSil
Started | 131
Completed | 131
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were treated with TachoSil and completed the study.
Arm/Group | TachoSil
Number analyzed (Participants) | 131
Age, Customized [Number; unit: participants]
  20-83 years | 131
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 131
Participants With Height From 152 to 190 Centimeter (cm) [Count of Participants; unit: Participants] | 131
Participants With Weight from 46.5 to 180 Kilogram (kg) [Count of Participants; unit: Participants] | 131

OUTCOME MEASURES:

1. Primary Outcome: Investigators Assessment of Tachosil
Description: Investigators were asked to evaluate the overall manageability and satisfaction with TachoSil in laparoscopic surgery. The overall manageability and satisfaction of TachoSil application was assessed using Likert scale. It is a 5-point scale, that ranges from 1-5, where 1=easy to use/satisfied to 5=difficult to use/not satisfied. Higher scores indicates difficulty and less satisfaction. The mean manageability satisfaction with the application of TachoSil were reported.
Time Frame: Post-surgery until hospital discharge (up to 13 days)
Population: The safety analysis set included all participants who were treated with TachoSil and completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TachoSil
Number analyzed (Participants) | 131
score on a scale
  Overall manageability | 1.91 (0.76)
  Overall satisfaction | 1.86 (0.80)

2. Secondary Outcome: Duration of Hospital Stay
Time Frame: From date of surgery until hospital discharge (up to 13 days)
Population: The safety analysis set included all participants who were treated with TachoSil and completed the study.
Measure: Median (Full Range); unit: days
Arm/Group | TachoSil
Number analyzed (Participants) | 131
days | 5 [3 to 13]

3. Secondary Outcome: Number of Participants With Pharmaco-economic Evaluation Based on Surgeon's Assessment
Description: Pharmaco-economic evaluation based on surgeon's assessment included surgery time, intensive care unit (ICU) time, total care time, and other advantages. Other advantages included reduced or no risk of secondary bleeding, and the easier application and manageability.
Time Frame: Intra-surgery and post-surgery until hospital discharge (up to 13 days)
Population: The safety analysis set included all participants who were treated with TachoSil and completed the study.
Measure: Number; unit: participants
Arm/Group | TachoSil
Number analyzed (Participants) | 131
participants
  Participants with reduction of surgery time | 10
  Participants with reduction of ICU time | 0
  Participants with reduction of total care time | 0
  Participants with other advantages | 8

4. Secondary Outcome: Number of Participants With Intra-operative and Post-operative Adverse Events (AEs)
Time Frame: Baseline up to 13 days
Population: The safety analysis set included all participants who were treated with TachoSil and completed the study.
Measure: Number; unit: participants
Arm/Group | TachoSil
Number analyzed (Participants) | 131
participants | 2

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) are AEs that started after the first application of open label study drug up to end of study (up to 13 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TachoSil
All-Cause Mortality (participants affected / at risk) | 0/131
Serious Adverse Events (participants affected / at risk) | 2/131
Other Adverse Events (participants affected / at risk) | 0/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TachoSil (N=131)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2015-08-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT02685007/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT02685007/SAP_001.pdf